CLINICAL TRIAL: NCT02757547
Title: Registered Electrical Sources for Effective TMS Treatment of Epilepsy
Brief Title: Transcranial Magnetic Stimulation for Epilepsy
Acronym: TMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to discontinue development of this investigational device.
Sponsor: Electrical Geodesics, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDEG150216
Record Dates: First submitted 2016-04-19; First posted 2016-05-02 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial magnetic stimulation - Placebo Arm (Placebo Comparator): A placebo TMS coil is used.
  Interventions: Device: Transcranial magnetic stimulation - Placebo Arm
- Transcranial magnetic stimulation - Active Arm (Active Comparator): An active TMS coil is used.
  Interventions: Device: Transcranial magnetic stimulation - Active Arm

INTERVENTIONS:
Device: Transcranial magnetic stimulation - Placebo Arm — Each seizure patient (subject) will receive 5 days in a row the placebo (sham) magnetic stimulation using the placebo (sham) coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total. The placebo coil produces the same noise and movement as an active coil, but doesn't deliver any magnetic stimulation.
  Arms: Transcranial magnetic stimulation - Placebo Arm
Device: Transcranial magnetic stimulation - Active Arm — Each seizure patient (subject) will receive 5 days in a row of active magnetic stimulation using the active TMS coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total.
  Other Names: STM9000 Transcranial Magnetic Stimulator
  Arms: Transcranial magnetic stimulation - Active Arm

SUMMARY:
The goal of the present clinical trial is to determine whether low frequency (0.5 Hz) rTMS can induce long term depression in epileptogenic cortex and thus suppress cortical excitability at the epileptic focus.

DETAILED DESCRIPTION:
Investigators propose a safety and feasibility trial for treating epilepsy (Transcranial Magnetic Stimulation for Epilepsy. Principal Investigator: Robert Fisher, MD, PhD, Stanford University). In this approach, the cortical source of epileptic discharges is first localized with dense array electroencephalography (256-channel dEEG). This localization is then registered with neuronavigator software to allow precise targeting with slow (0. 5 Hz) repetitive Transcranial Magnetic Stimulation (rTMS) with the STM9000. The purpose in the feasibility study is to introduce Long Term Depression (LTD) of the seizure onset zone in order to reduce epileptiform discharges. The goal in the future pivotal trial will be to extend this approach to suppress seizures. The funds for this trial are provided by Stanford University. A loan of dEEG equipment and consulting are provided by Electrical Geodesics, Inc. (EGI). EGI seeks FDA's approval for this trial. EGI is the manufacturer of the dEEG system (GES 400) and the US distributor of the EB Neuro STM9000 rTMS system (manufactured in Italy by EB Neuro, S.p.A.).

The eventual goal will be a pivotal trial for a de novo 510k for dEEG-guided rTMS for suppressing epileptic seizures. The more limited goal of suppressing epileptic discharges (spikes) will allow careful evaluation of safety while demonstrating feasibility of the therapeutic action. In preparing this request, the investigators have studied the guidance on the special controls described for rTMS in the FDA Class II Special Controls Guidance Document: Repetitive Transcranial Magnetic Stimulation (rTMS) Systems, Document issued on: July 26, 2011. In addition, because patients with epilepsy are at particular risk of seizures that may be induced or exacerbated by rTMS, investigators also address the unique risks of this population, the existing evidence on safety and efficacy of rTMS treatment of the epileptic focus, and the mitigation the investigators propose to minimize the risks.

EGI has received an IDE for a safety and feasibility trial for treating epileptic discharges with a different method and device, the Geodesic Transcranial Electrical Neuromodulation (GTEN 100) system. The primary difference in the present proposal is the use of rTMS (instead of the GTEN 100) to induce long term depression and thus suppression of the cortical excitability at the epileptic focus. Dr. Robert Fisher, the Principal Investigator on this project, is EGI's unpaid consultant. Dr. Fisher has received an IRB approval at Stanford University Hospital for the larger study with this title for 10 patients with dEEG-guided rTMS treatment of focal epilepsy with the GES 400 and STM9000. The present trial is a safety and feasibility study with 10 patients that will be conducted with an informed consent form that is now specific to this safety and feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. Failure of adequate seizure control with prior use of at least 2 anti-seizure drugs.
2. at least one clearly identified and localizable likely seizure onset focus, as defined by the discharges (typically epileptiform spikes) and as identified by dEEG assessment through one or more routine clinical dEEG evaluations. This focus must be 2 to 3 cm from the head surface (to be reachable by TMS). Where multiple spike foci are present and meet these criteria, then the focus with either clinically relevant symptoms or the most spikes (or both) will be chosen as the target for treatment.
3. two or more partial seizures, with or without secondary generalization, in the last month, but less than 10 seizures per day.
4. Anti-seizure drug regimen has remained unchanged for the month before study entry, and there is reasonable likelihood of stability for the duration of the study, with the exception of allowing short-term rescue medications, such as lorazepam.
5. a history of epilepsy for at least 2 years.
6. age of 22 years and older.

Exclusion Criteria:

1. If of childbearing potential, the patient must agree to use an effective method of birth control during the study and cease participation if pregnant.
2. Nursing mothers are excluded.
3. A history or condition of progressive brain disorders, serious systemic diseases, symptomatic cerebrovascular disease, cardiac disease, or alcohol abuse. Special conditions, for example, non-malignant brain tumors and vascular malformations, can be considered for entry on a case-by-case basis. Patients are not excluded on the basis of previous psychiatric hospitalizations or suicide attempts.
4. A history or condition of (generalized) status epilepticus or psychogenic seizures.
5. Presence of a cardiac pacemaker, vagus nerve stimulator, or metal implantation in the body (other than the teeth) including neurostimulators, cochlear implants, and implanted medication pumps.
6. Previous surgery involving opening the skull.
7. Unable to express presence of pain or discomfort.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fisher, Ph.D., Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects participating in the study will undergo both arms. Subjects will first complete the Placebo Arm and then will complete the Active Arm.
Groups:
- TMS Placebo Arm Followed by TMS Active Arm: A placebo TMS coil is used for the Placebo Arm
  Transcranial magnetic stimulation - Placebo Arm: Each seizure patient (subject) will receive 5 days in a row the placebo (sham) magnetic stimulation using the placebo (sham) coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total. The placebo coil produces the same noise and movement as an active coil, but doesn't deliver any magnetic stimulation.
  TMS Active Arm:
  An active TMS coil is used. Transcranial magnetic stimulation - Active Arm: Each seizure patient (subject) will receive 5 days in a row of active magnetic stimulation using the active TMS coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total.
Period: Overall Study
Arm/Group | TMS Placebo Arm Followed by TMS Active Arm
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- TMS - Placebo Arm Followed by Active Arm: A placebo TMS coil is used for the Placebo Arm:
  Transcranial magnetic stimulation - Placebo Arm: Each seizure patient (subject) will receive 5 days in a row the placebo (sham) magnetic stimulation using the placebo (sham) coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total. The placebo coil produces the same noise and movement as an active coil, but doesn't deliver any magnetic stimulation.
  An active TMS coil is used for the Active Arm:
  Transcranial magnetic stimulation - Active Arm: Each seizure patient (subject) will receive 5 days in a row of active magnetic stimulation using the active TMS coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total.
Arm/Group | TMS - Placebo Arm Followed by Active Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Suppression of Seizure Frequency
Description: The primary outcome was determined to be measured by the reduction in seizure frequency compared to baseline.
Time Frame: Placebo compared to Active
Population: The study was initiated by Electrical Geodesics Inc. At the time of the acquisition it was determined that the study was not in compliance with the regulations and/or GCP. There was no protocol, no statistical analysis plan, no case report forms and no data was monitored or collected therefore, no statistical analysis could be performed.
Groups:
- TMS - Placebo Arm Followed by Active Arm: A placebo TMS coil is used.
  Transcranial magnetic stimulation - Placebo Arm: Each seizure patient (subject) will receive 5 days in a row the placebo (sham) magnetic stimulation using the placebo (sham) coil of the STM9000 Transcranial Magnetic Stimulator. This involves magnetic stimulation at 90% of the resting motor threshold at 1 Hz in three 500-pulse blocks, separated by 10-minute breaks for 1500 pulses total. The placebo coil produces the same noise and movement as an active coil, but doesn't deliver any magnetic stimulation.
Arm/Group | TMS - Placebo Arm Followed by Active Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Investigator observed subjects for adverse events over the course of the study from enrollment to the last follow-up (e.g., 9 months)
Arm/Group | Transcranial Magnetic Stimulation - Placebo Arm | Transcranial Magnetic Stimulation - Active Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT02757547/Prot_SAP_000.pdf